CLINICAL TRIAL: NCT02233192
Title: PrEPception: Expanding Assisted Reproductive Options for Serodiscordant Couples
Status: Completed | Type: Observational
Sponsor: Boston Medical Center (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: H-33071
Record Dates: First submitted 2014-08-19; First posted 2014-09-08 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: PrEP for Conception Purposes
Keywords: PrEP; conception; HIV; serodiscordant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — To measure levels of PrEP to assess medication adherence, approximately 4ml of blood will be drawn on female participants (2 tests total for the study period). One dried blood spot will be collected after steady state tenofovir (approximately one month after beginning PrEP) is reached and one at the time a pregnancy is confirmed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to observe patient response to current clinical practice utilizing TRUVADA (emtricitabine and tenofovir disoproxil fumarate) for Pre-Exposure Prophylaxis (PrEP) amongst HIV serodiscordant couples desiring to conceive across four U.S. cities that are currently offering this method as standard of care. This study is an observational cohort study, which will test the feasibility and acceptability of PrEP for conception, while examining the challenges and generalizability of this current medical practice. The CDC recently released formal clinical practice guidelines for the use of PrEP in the United States. For high-risk serodiscordant heterosexual couples using PrEP during conception, the guidelines state, "PrEP use periconception and during pregnancy by the uninfected partner may offer an additional tool to reduce the risk of sexual HIV acquisition. Both the FDA labeling information and the perinatal antiretroviral treatment guidelines permit this use" (CDC 2014).

DETAILED DESCRIPTION:
Based on CDC's guidance on PrEP as well as results of randomized controlled trials, the U.S. Food and Drug Administration (FDA) approved this daily medication (comprised of one pill) to reduce the risk of sexually acquired HIV in adults at high risk. Other medical practices to avoid transmission within this population include assisted reproductive technologies such as sperm washing (or donated sperm) coupled with in vitro fertilization, intracytoplasmic sperm injection (an in vitro procedure where a single sperm is injected directly into an egg), and intrauterine insemination (placing the sperm directly into the uterus). However, these methods are costly and often regionally scarce. PrEP is more accessible and a less expensive option for couples. When used consistently and as prescribed, PrEP has shown to significantly reduce the risk of HIV infection among adult men and women. However, risk reduction counseling and clinical monitoring are necessary for its effective implementation. Therefore, beyond efficacy trials, it is important to conduct additional studies of pre-exposure prophylaxis to observe what factors make PrEP feasible and acceptable to couples, as well as identify other factors that impact level of adherence. The study will take place in four U.S. cities: Boston, Baltimore, Philadelphia, and San Francisco and will involve couples who have chosen to begin PrEP for conception as part of their clinical care after receiving preconception counseling and reviewing their options with their health care provider.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 to 40 years
* In relationship with HIV-positive male
* Chosen to take PrEP for conception after completing counseling with health care provider

Exclusion Criteria:

* HIV-positive
* In relationship with HIV-negative female
* Partner has chosen to take PrEP for conception after completing counseling with health care provider

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will take place in teaching hospitals in four U.S. cities: Boston, Baltimore, Philadelphia, and San Francisco and will involve couples who have chosen to begin PrEP for conception as part of their clinical care after receiving preconception counseling and reviewing their options with their health care provider.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Change in PrEP adherence levels throughout regimen | Monthly; participants will be followed for the duration of trying to conceive, an expected average of 1 year
  Adherence will be measured in two ways: (1) Dried blood spots (DBS) to measure drug level two times, once after the woman has been taking the drug for one month and once when pregnancy is confirmed. We will perform unadjusted, bivariate analyses comparing participants below and equal to the drug level threshold for daily dosing using a one sample t-test for normally distributed continuous or ordinal variables on adherence. We will also perform a paired t-test for measuring the difference, if any, between the two adherence tests at the different time points for each individual. Adherence will also be measured through (2) participant self-report via a continuous variable of number of doses missed in the past month. We will perform unadjusted, bivariate analyses comparing the observed participant self-reported adherence levels to the gold standard of ≥95% self-reported adherence using a one-sample t test of means for normally distributed continuous or ordinal variables.
Change in condom use and sexual practice over time | Participants will be followed for the duration of trying to conceive, an expected average of 1 year
  Condom use will be measured through participant self-report on number of times a condom was used during the past month compared to the number of times the participant had sexual intercourse with his/her partner or other individuals in the past month. We will perform unadjusted bivariate analyses comparing the observed participants in a one-sample student's t-test for normally distributed variables on condom use or a paired t-test for measuring the difference between two variables at different time points for the same subject (i.e. at baseline and at end-line evaluation). For a non-normal distribution, we will use the non-parametric equivalent such as Sign or Wilcoxon Signed rank test for a symmetric distribution.
Change in number of couples who complete a clinical protocol for PrEP compared to the total number of couples that initiate PrEP | Monthly; participants will be followed for the duration of trying to conceive, an expected average of 1 year
  We will quantify this outcome measure by examining the number of couples who complete a clinical protocol for PrEP compared to the total number of couples that initiate PrEP, while examining other variables that could make the two groups statistically different. We will perform unadjusted bivariate analyses comparing the number of couples that complete the clinical protocol and those who withdraw or become ineligible throughout the duration of the study. We will use a one-way ANOVA or Kruskal-Wallis non-parametric test for continuous variables with two or more categories such as those that complete the protocol versus those that withdraw from PrEP versus those that become ineligible. We will perform a two-sample test of means to compare the overall categories of those that complete the protocol versus those that do not complete the protocol and create cross-tabulations with chi-square and Fisher's exact tests.
Change in beliefs and sexual behavior at different time points for the same subject | Monthly; participants will be followed for the duration of trying to conceive, an expected average of 1 year
  For this outcome measure, we will perform unadjusted bivariate analyses in a paired t-test for measuring the difference in beliefs and sexual behavior at different time points for the same subject. For a non-normal distribution, we will use the non-parametric equivalent such as Sign or Wilcoxon Signed rank test for a symmetric distribution.

SECONDARY OUTCOMES:
Changes in creatinine clearance from the baseline compared to creatinine clearance at the conclusion of PrEP for the same subject | Participants will be followed for the duration of trying to conceive, an expected average of 1 year
  To assess renal toxicities, we will perform unadjusted bivariate analyses in a paired t-test for measuring the difference of creatinine clearance from the baseline compared to creatinine clearance at the conclusion of PrEP for the same subject. For a non-normal distribution, we will use the non-parametric equivalent such as Sign or Wilcoxon Signed rank test for a symmetric distribution. We will also report on basic drug side effects, while summarizing other self-reported effects of PrEP.
Measuring the rates of teratogenicity as compared to the general population as determined by medical record review | 1 year
  We will perform unadjusted bivariate analyses in a two-sample test of means to compare rates of teratogenicity of newborns with HIV-negative females using PrEP as compared to rates of birth defects within the general population in similar age group women.
HIV transmission rates | Participants will be followed for the duration of trying to conceive, an expected average of 1 year
  For this outcome measure, we will report descriptively on whether there is a transmission or not within the observed participants taking PrEP for conception purposes.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Sullivan, MD, Principal Investigator — Boston University
Locations (4):
- United States (4):
  - Northwestern University, Chicago, Illinois
  - The Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Boston University Medical Center, Boston, Massachusetts
  - Drexel University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No